CLINICAL TRIAL: NCT00813072
Title: A Randomized Phase II Study of PEP02, Irinotecan or Docetaxel as a Second Line Therapy in Patients With Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Study of PEP02, Irinotecan or Docetaxel in Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaEngine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEP0206; EudraCT number: 2006-006452-35
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-03

CONDITIONS: Stomach Neoplasms; Esophageal Neoplasms
Keywords: Gastric Cancer; Stomach Cancer; Gastroesophageal; Gastroesophageal Junction; Esophageal Cancer; phase II; PEP02; randomization; randomisation; adenocarcinoma; locally advanced; metastatic; simon's two
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Adenocarcinoma; Neoplasm Metastasis | interventions — Irinotecan; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1. PEP02 (Experimental): liposome irinotecan
  Interventions: Drug: PEP02
- 2. irinotecan (Active Comparator)
  Interventions: Drug: irinotecan
- 3. docetaxel (Active Comparator)
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: PEP02 — 120 mg/m2, IV infusion for 90 minutes on day 1 of each 21 day as a treatment cycle.
  Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: liposome irinotecan
  Arms: 1. PEP02
Drug: irinotecan — 300 mg/m2, IV infusion on day 1 of each 21 day as a treatment cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Campto
  Arms: 2. irinotecan
Drug: docetaxel — 75 mg/m2, IV infusion for 60 minutes on day 1 of each 21 day as a treatment cycle.
  Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Taxetere
  Arms: 3. docetaxel

SUMMARY:
The purpose of this study is to assess objective tumor response in the single agent treatment of PEP02, irinotecan, or docetaxel for locally advanced or metastatic gastric or gastroesophageal junction adenocarcinoma

DETAILED DESCRIPTION:
Palliative chemotherapy has been shown to improve survival compared with best supportive care alone in patients with unresectable or recurrent gastric cancer. There is no standard second-line chemotherapy for advanced gastric cancer and no randomized-controlled trial data suggest a benefit of second-line chemotherapy compared with supportive care alone. Response rates of second-line therapy in phase II trials are similar to those seen for other cancers that are more commonly retreated. Combination therapy may achieve higher response rates than single agents, however, the survival outcome are the same. In addition, data suggest that patients may obtain symptomatic benefits from second-line therapy. In comparison to the toxicity profile of single agent with combination regimen, patients are more tolerable to single agent therapy than combination.

Based on the previous clinical experience in second line chemotherapy of advanced gastric cancer, the single agent of PEP02, irinotecan and docetaxel are selected as the regimens for this randomized phase II study. The efficacy and toxicity outcome of the three-arm design will be a valuable reference for future combination therapy or phase III study design.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced (unresectable) or metastatic adenocarcinoma of gastric or gastroesophageal junction
* Failed to only one systemic chemotherapy for locally advanced or metastatic disease, including patients whose diseases recur within 6 months after (neo)adjuvant chemotherapy. Chemotherapy administered with concurrent radiotherapy is NOT considered as systemic chemotherapy.
* Have at least one measurable lesion according to the RECIST criteria
* Aged above or equal to 18 years, at the time of acquisition of informed consent
* With ECOG performance status 0, 1, or 2
* Life expectancy equal to or more than 3 months
* With adequate organ and marrow function as defined below:
* With ability to understand and the willingness to sign a written Informed Consent Form

Exclusion Criteria:

* Had systemic chemotherapy within 3 weeks before the commencement of study treatment
* Had radiotherapy within 4 weeks before the commencement of study treatment
* With known brain metastasis
* With active multiple cancers or had treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer
* With prior irinotecan or taxane (paclitaxel, docetaxel) treatment
* Have received irradiation affecting > 30% of the active bone marrow
* Had major surgery within 4 weeks of the start of study treatment (laparotomy, line placement is not considered major surgery)
* Have not recovered from prior treatments
* With preexisting peripheral neuropathy > grade 2
* With history of allergic reaction to liposome product or other drugs formulated with polysorbate
* With uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, active gastrointestinal bleeding, watery stools, central nervous system disorders or psychiatric illness/social situation that would limit compliance with study requirements or judged to be ineligible for the study by the investigator
* Have received any investigational agents within 3 weeks preceding the start of study treatment
* Pregnant or breastfeeding females (a pregnancy test must be performed on all female patients who are of child-bearing potential before entering the study, and the result must be negative)
* With intestinal obstruction
* Have received St. John's Wort, CYP3A4 inducing anticonvulsants (phenytoin, phenobarbital, and carbamazepine), rifampin and rifabutin within two weeks, or ketoconazole, itraconazole, troleandomycin, erythromycin, diltiazem and verapamil within one week before the administration of study medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2007-11; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
objective tumor response

SECONDARY OUTCOMES:
progression-free survival, duration of tumor response, time to progression, time to treatment failure, disease control rate, 1-year survival rate,and overall survival; pharmacokinetics and pharmacogenetics of PEP02 and irinotecan

CONTACTS AND LOCATIONS:
Overall Officials: David Cunningham, Principal Investigator — The Royal Marsden Hospital, London & Surrey, UK
Locations (22):
- Bosnia and Herzegovina (2):
  - Clinical Hospital Mostar, Mostar
  - Clinical Centre University of Sarajevo, Sarajevo
- Croatia (3):
  - University Hospital Centre Rijeka, Rijeka
  - University Hospital Centre Dubrava, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- South Korea (3):
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - National Cancer Center, Seoul
- Spain (4):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
- Taiwan (5):
  - Chang Gung Memorial Hospital - Chiayi, Chiayi City
  - Chang Gung Memorial Hospital - LinKou, Linkou District
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
- United Kingdom (5):
  - Addenbrookes Hospital Oncology Center, Cambridge
  - Guy's & St Thomas' NHS Foundation Trust, London
  - Kent Oncology Centre, Maidstone Hospital, Maidstone
  - Southampton University Hospital, Southampton
  - The Royal Marsden Hospital, Surrey

REFERENCES:
- [Derived] Roy AC, Park SR, Cunningham D, Kang YK, Chao Y, Chen LT, Rees C, Lim HY, Tabernero J, Ramos FJ, Kujundzic M, Cardic MB, Yeh CG, de Gramont A. A randomized phase II study of PEP02 (MM-398), irinotecan or docetaxel as a second-line therapy in patients with locally advanced or metastatic gastric or gastro-oesophageal junction adenocarcinoma. Ann Oncol. 2013 Jun;24(6):1567-73. doi: 10.1093/annonc/mdt002. Epub 2013 Feb 13. PMID 23406728